CLINICAL TRIAL: NCT04793295
Title: A Phase I, Open-Label, Four-Part, Single-Sequence Study to Investigate Drug-Drug Interaction Between MT-7117 and Test Drugs in Healthy Subjects
Brief Title: Study to Investigate Drug-Drug Interaction Between MT-7117 and Test Drugs in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MT-7117-Z-102
Record Dates: First submitted 2021-03-10; First posted 2021-03-11 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MT-7117 Drug-drug interaction with test drug 1 and test drug 2 (Experimental)
  Interventions: Drug: MT-7117
- MT-7117 Drug-drug interaction with test drug 3 and test drug 4 (Experimental)
  Interventions: Drug: MT-7117
- MT-7117 Drug-drug interaction with test drug 5 and test drug 6 (Experimental)
  Interventions: Drug: MT-7117
- MT-7117 Drug-drug interaction with test drug 7 (Experimental)
  Interventions: Drug: MT-7117

INTERVENTIONS:
Drug: MT-7117 — MT-7117
  Other Names: Dersimelagon

SUMMARY:
Study is to investigate drug levels in the blood after taking single or multiple doses of the study drug, MT-7117, in healthy adults when taken together with another drug. This study will also look at the safety and the body's ability to tolerate MT-7117

ELIGIBILITY:
Inclusion Criteria: Subjects will be eligible for inclusion in the study if they meet all of the following criteria:

1. Able and willing to provide written informed consent to participate in this study after reading the participant information sheet and Informed Consent Form (ICF) and having the opportunity to discuss the study with the Investigator or designee.
2. Male and female subjects, self-reporting as white, 18-55 years of age, inclusive, at the time of signing the ICF.
3. Subjects must weigh at least 50 kg (110 pounds) and have a body mass index 18-30 kg/m2, inclusive, at Screening and on Day -1.
4. Female subjects must not be lactating, and women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test within 24 hours prior to receiving the first dose of IMP or IMP Test Products.
5. Female subjects of childbearing potential and male subjects with a partner of childbearing potential must agree to use 2 effective methods of contraception (in female subjects, one method must be highly effective). Full details of contraception in Section 4.6.5.
6. In the Investigator's opinion, the subject must be able to understand the nature of the study and any risks involved in participation and be willing to cooperate and comply with the protocol restrictions and requirements.

Exclusion Criteria: Any subject meeting any of the following criteria will not qualify for enrolment in the study:

1. Presence or history of any hepatobiliary disease at Screening, determined clinically significant by the Investigator after discussion with the Sponsor's Responsible Physician. Current, or history of, clinically significant (in the opinion of the Investigator AND Sponsor's Responsible Physician) neurological conditions, endocrine, thyroid, respiratory, gastrointestinal, renal, or cardiovascular disease, or history (within the last 2 years) of any clinically significant psychiatric/psychotic illness disorder (including anxiety, depression, and reactive depression).
2. Clinically relevant abnormal medical history, physical findings, or laboratory values at Screening or Day-1 that could interfere with the objectives of the study or the safety of the subjects, in the opinion of the Investigator.
3. A history of gastrointestinal surgery known to affect the absorption, metabolism, or excretion of the IMP or IMP Test Products such as bariatric surgery or removal of part of the bowel. A history of appendicectomy and hernia repair/herniorrhaphy/hernioplasty is permitted for inclusion in the study.
4. Family history of long or short QT syndrome, hypokalemia, syncope, or Torsades de Pointes.
5. Clinically significant 12-lead electrocardiogram (ECG) abnormalities, including subjects with corrected QC interval (QTc) using Fridericia's formula >450 ms (male) and >470 ms (female), at Screening or Day -1. A repeat assessment is allowed at each visit. If the repeat measurement is in range, the subject may be included.
6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) 1.5 the upper limit of normal (ULN) reference range, or bilirubin ≥ 1.5 ULN at screening or Day-1. A repeat assessment is allowed at each visit. If the repeat measurement is in range, the subject may be included.
7. Systolic blood pressure outside the range of 90-145 mmHg, diastolic blood pressure outside the range of 50-95 mmHg, or pulse rate outside the range of 50-100 bpm, taken in the supine position at Screening or Day -1. A repeat assessment is allowed at each visit. If the repeat measurement is in range, the subject may be included.
8. Receipt of any prescribed of nonprescribed systemic or topical medication within 30 days (or, if relevant, 5 half-lives, whichever is longer) prior to the first dose of study drugs unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise subject safety.

   1. Occasional use of paracetamol (acetaminophen) for mild analgesia is permitted.
   2. Vitamins and herbal supplements are not permitted 14 days prior to dosing
9. Presence or history of severe adverse reaction or allergy to food or any drug or excipient or other allergy that is of clinical significance to the study drugs.
10. Previous receipt of MT-7117.
11. First-degree relative with a history of familial melanoma.
12. Previous use of afamelanotide or melanotan.
13. Female subjects planning to donate eggs (during the study and for 3 months after the last visit).
14. Positive test for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV) 1 or HIV 2 antibodies at Screening.
15. Presence or history of drug abuse (as defined by Diagnostic and Statistical Manual of Mental Disorders criteria), or a positive urine test for drugs of abuse at Screening or Day -1.
16. Presence or history (in the last 2 years) of alcohol abuse or excessive alcohol consumption, defined as subjects who regularly, or on average, drink more than 21 units (168 g) for males or 14 units (112 g) for females, of alcohol per week (1 unit is equivalent to 8 g of alcohol).
17. Use of tobacco or nicotine-containing products (snuff, chewing tobacco, cigarettes, cigars, pipes, e-cigarettes, or nicotine replacement products) within 3 months prior to dosing, or a positive urine cotinine test at Screening or Day -1.
18. Consumption of food or drink containing oranges, grapefruit, liquorice, or cranberry within the 7 days prior to the first dose of study drug.
19. Subjects who are not willing to abstain from consumption of caffeine and methylxanthine (e.g., coffee, tea, cola, energy drinks, or chocolates) in the 48 hours before Day -1 until completion of the post-treatment assessments and in the 48 hours before the Follow-up/End of Study Visit.
20. Donation of 1 or more units of blood (450 mL) in the 3 months prior to Screening, plasma in the 7 days prior to Screening, platelets in the 6 weeks prior to Screening, or the intention to donate blood within 3 months after the last scheduled visit.
21. Heavy physical training, labor, or excessive exercise (e.g., long-distance running, weightlifting, or any physical activity to which the subject is not accustomed) from 3 days before the administration of study drugs.
22. Participation in more than 3 clinical studies* involving administration of an IMP in the previous year, or any study* involving administration of an IMP within 8 weeks (or, if relevant, 5 half-lives, whichever is longer) prior to the first dose of study drug.

    *Disregarding any study Follow-up Periods.
23. Subjects with the presence of a skin lesion suspicious for dysplastic nevus or a history of histologically proven dysplastic nevus.
24. Subjects who have any active malignancy (including melanoma) or history of significant malignancy (including melanoma).
25. Subjects who have had Coronavirus Disease 2019 (COVID-19) in the 3 months prior to Screening; or suspected active COVID-19 infection, a positive COVID-19 test, contact with an individual with known COVID-19, or travel to an area with a high risk of COVID-19 infection within 14 days of Screening.
26. Subjects that test positive for COVID-19 at Screening (Parts 3 and 4) or Day -1 (Parts 1-4).
27. Subjects who have received a COVID-19 vaccination within 14 days of Day 1. COVID-19 vaccination is not permitted during the study. Subjects may not take part in the study if they have started but not completed a COVID-19 vaccination course at the time of Screening or Day -1.
28. Subjects who have a history of major surgery within 3 months of Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products in the absence and presence of MT-7117 (Parts 1, 2, and 3) and MT-7117 in the absence and presence of test drug 7 (Part 4)
Area under the plasma concentration-time curve (AUC) from time zero to infinity (AUC0-∞) | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products in the absence and presence of MT-7117 (Parts 1, 2, and 3) and MT-7117 in the absence and presence of test drug 7 (Part 4)
AUC from time zero to the last measurable concentration (AUC0-last) | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products in the absence and presence of MT-7117 (Parts 1, 2, and 3) and MT-7117 in the absence and presence of test drug 7 (Part 4)

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (tmax) | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products in the absence and presence of MT-7117 (Parts 1, 2, and 3) and MT-7117 in the absence and presence of test drug 7 (Part 4)
t1/2 | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products in the absence and presence of MT-7117 (Parts 1, 2, and 3) and MT-7117 in the absence and presence of test drug 7 (Part 4)
Apparent oral clearance | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products in the absence and presence of MT-7117 (Parts 1, 2, and 3) and MT-7117 in the absence and presence of test drug 7 (Part 4)
Apparent volume of distribution during the terminal phase after oral administration | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products in the absence and presence of MT-7117 (Parts 1, 2, and 3) and MT-7117 in the absence and presence of test drug 7 (Part 4)
Cmax | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products metabolites in the absence and presence of MT-7117 (Parts 1, 2, and 3)
tmax | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products metabolites in the absence and presence of MT-7117 (Parts 1, 2, and 3)
t1/2 | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products metabolites in the absence and presence of MT-7117 (Parts 1, 2, and 3)
AUC0-last | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products metabolites in the absence and presence of MT-7117 (Parts 1, 2, and 3)
AUC0-∞ | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
  PK parameters of IMP Test Products metabolites in the absence and presence of MT-7117 (Parts 1, 2, and 3)
MT-7117 concentrations in plasma | Part 1 Day 1 to Day 19, Part 2 Day 1 to Day 15, Part 3 Day 1 to Day 17, Part 4 Day 1 to Day 13
Safety and tolerability as measured by incidence of adverse events | Part 1 Day -1 to Day 25, Part 2 Day -1 to Day 21, Part 3 Day -1 to Day 23, Part 4 Day -1 to Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (2):
- United States (2):
  - Advanced Pharma CR, LLC, Miami, Florida
  - Worldwide Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogasawara A, Ide R, Inoue S, Tsuda M, Teng R. Assessment of Potential Drug-Drug Interactions for Novel Oral Melanocortin-1 Receptor Agonist Dersimelagon. Pharmacol Res Perspect. 2025 Feb;13(1):e70069. doi: 10.1002/prp2.70069. PMID 39887900